CLINICAL TRIAL: NCT05279131
Title: A Phase 3, Multicenter, Open-label, Single-arm Study to Evaluate the Safety and Tolerability of Tirbanibulin Ointment 1% Applied to a Field of Approximately 100 cm2 on the Face or Balding Scalp in Adult Patients With Actinic Keratosis
Brief Title: A Study to Evaluate the Safety and Tolerability of Tirbanibulin Ointment 1% in Adult Participants With Actinic Keratosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-14867-32
Record Dates: First submitted 2022-03-01; First posted 2022-03-15 (Actual); Results first posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-12

CONDITIONS: Keratosis, Actinic
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tirbanibulin (Klisyri®) (Experimental): Participants will apply tirbanibulin ointment 1% once daily for 5 days beginning Day 1. Participants will be evaluated for safety, tolerability, and the presence of Actinic Keratosis (AK) lesions in the treatment field (TF) until completion of the response assessment period at Day 57.
  Interventions: Drug: Tirbanibulin ointment 1%

INTERVENTIONS:
Drug: Tirbanibulin ointment 1% — Applied topically for 5 days over a field of approximately 100 cm^2 on the face or balding scalp with AK.

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability and treatment effect of tirbanibulin ointment 1% when applied to a field of approximately 100 cm^2 on the face or balding scalp.

ELIGIBILITY:
Inclusion Criteria:

* Having a treatment field (TF) on the face or balding scalp (excluding lips, eyelids, and inside nostrils and ears) that measures approximately 100 cm^2 (eg, mid face) and contains 4 to 12 clinically typical, visible, and discrete actinic keratosis (AK) lesions within the TF
* Willing to avoid excessive sunlight or ultraviolet (UV) light exposure, including the use of tanning beds, to the face or scalp during the study
* Ability to understand the purpose and risks of the trial, willingness and ability to comply with the protocol, and provided written informed consent in accordance with institutional and regulatory guidelines

Exclusion Criteria:

* Presence in the TF of

  1. Clinically atypical and/or rapidly changing AK lesions in the TF
  2. Hyperkeratotic or hypertrophic lesions, recalcitrant disease (had cryosurgery on 2 previous occasions) and/or cutaneous horn
  3. Confluent AK lesions (ie, non-discrete lesions defined as per inclusion criteria)
  4. History of invasive squamous cell carcinoma (SCC), Bowen's disease, basal cell carcinoma (BCC), or other malignant tumors in the TF
  5. Any other dermatological disease that causes difficulty with examination
* Previous treatment with tirbanibulin ointment 1%.
* Anticipated need for inpatient hospitalization or inpatient surgery from Day 1 to Day 57
* Treatment with 5-fluorouracil, imiquimod, ingenol mebutate, diclofenac, photodynamic therapy, or other treatments for AK within the TF or within 2 cm of the TF, within 8 weeks prior to the Screening visit
* Use of systemic retinoids (eg, isotretinoin, acitretin, bexarotene) within 6 months prior to the Screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Almirall Investigation Site 7, Hot Springs, Arkansas
  - Almirall Investigation Site 6, Encinitas, California
  - Almirall Investigation Site 3, Sweetwater, Florida
  - Almirall Investigation Site 5, Rolling Meadows, Illinois
  - Almirall Investigation Site 4, Austin, Texas
  - Almirall Investigational Site 1, College Station, Texas
  - Almirall Investigation Site 2, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 20 sites in the United States from 28 June 2022 to 28 December 2022.
Pre-assignment Details: A total 105 participants were enrolled in the study to receive study treatment. At least 50 percent (%) of the participants were 65 years old (65%) and 71 participants were treated on the face and 34 participants on the scalp. The study consisted of a 4-week (28-day) Screening Period, a 5-day Treatment Period, and a Response Assessment Period of approximately 7 weeks.
Groups:
- Tirbanibulin (Klisyri®): Participants applied tirbanibulin ointment 1% topically once daily on Day 1 for 5 days over a field of approximately 100 square centimeters (cm^2) on the face or balding scalp with Actinic Keratosis (AK).
Period: Overall Study
Arm/Group | Tirbanibulin (Klisyri®)
Started | 105
Completed | 102
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Death | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all enrolled participants who received at least 1 dose of the study drug.
Groups:
- Tirbanibulin (Klisyri®): Participants applied tirbanibulin ointment 1% topically once daily on Day 1 for 5 days over a field of approximately 100 cm^2 on the face or balding scalp with AK.
Arm/Group | Tirbanibulin (Klisyri®)
Number analyzed (Participants) | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (8.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 98
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 105
  More than one race | 0
  Unknown or Not Reported | 0
Number of AK lesions at baseline [Mean (Standard Deviation); unit: Number of AK lesions] | 7.7 (2.72)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Categorized by Local Tolerability Score by Visit for Each Individual Signs (Erythema, Flaking/Scaling, Crusting, Swelling, Vesiculation/Pustulation, and Erosion/Ulceration) at Day 5
Description: Local tolerability score was evaluated by investigator in terms of presence and absence of erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration signs and its severity in the areas of body where medication was applied. These symptoms were assessed by using a 4 - point grade scale of 0 - 3, where a score of 0=absent, 1=mild (slightly, barely perceptible), 2=moderate (distinct presence), and 3=severe (marked, intense). The higher score indicates severe symptoms. Number of participants categorized by local tolerability score by visit for each individual signs (erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration) at Day 5 were reported.
Time Frame: Baseline, Day 5
Population: The safety population included all enrolled participants who received at least 1 dose of the study drug. Here, "Number analyzed" signifies participants who were evaluated at specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Tirbanibulin (Klisyri®)
Number analyzed (Participants) | 105
Participants
  Baseline: Erythema: Grade 0 | 81
  Baseline: Erythema: Grade 1 | 19
  Baseline: Erythema: Grade 2 | 5
  Baseline: Erythema: Grade 3 | 0
  At Day 5: Erythema: number analyzed (Participants) | 101
  At Day 5: Erythema: Grade 0 | 13
  At Day 5: Erythema: Grade 1 | 41
  At Day 5: Erythema: Grade 2 | 44
  At Day 5: Erythema: Grade 3 | 3
  Baseline: Flaking/Scaling: Grade 0 | 84
  Baseline: Flaking/Scaling: Grade 1 | 17
  Baseline: Flaking/Scaling: Grade 2 | 4
  Baseline: Flaking/Scaling: Grade 3 | 0
  At Day 5: Flaking/Scaling: number analyzed (Participants) | 101
  At Day 5: Flaking/Scaling: Grade 0 | 44
  At Day 5: Flaking/Scaling: Grade 1 | 38
  At Day 5: Flaking/Scaling: Grade 2 | 19
  At Day 5: Flaking/Scaling: Grade 3 | 0
  Baseline: Crusting: Grade 0 | 103
  Baseline: Crusting: Grade 1 | 2
  Baseline: Crusting: Grade 2 | 0
  Baseline: Crusting: Grade 3 | 0
  At Day 5: Crusting: number analyzed (Participants) | 101
  At Day 5: Crusting: Grade 0 | 90
  At Day 5: Crusting: Grade 1 | 9
  At Day 5: Crusting: Grade 2 | 2
  At Day 5: Crusting: Grade 3 | 0
  Baseline: Swelling: Grade 0 | 105
  Baseline: Swelling: Grade 1 | 0
  Baseline: Swelling: Grade 2 | 0
  Baseline: Swelling: Grade 3 | 0
  At Day 5: Swelling: number analyzed (Participants) | 101
  At Day 5: Swelling: Grade 0 | 73
  At Day 5: Swelling: Grade 1 | 25
  At Day 5: Swelling: Grade 2 | 3
  At Day 5: Swelling: Grade 3 | 0
  Baseline: Vesiculation/Pustulation: Grade 0 | 105
  Baseline: Vesiculation/Pustulation: Grade 1 | 0
  Baseline: Vesiculation/Pustulation: Grade 2 | 0
  Baseline: Vesiculation/Pustulation: Grade 3 | 0
  At Day 5: Vesiculation/Pustulation: number analyzed (Participants) | 101
  At Day 5: Vesiculation/Pustulation: Grade 0 | 98
  At Day 5: Vesiculation/Pustulation: Grade 1 | 3
  At Day 5: Vesiculation/Pustulation: Grade 2 | 0
  At Day 5: Vesiculation/Pustulation: Grade 3 | 0
  Baseline: Erosion/Ulceration: Grade 0 | 105
  Baseline: Erosion/Ulceration: Grade 1 | 0
  Baseline: Erosion/Ulceration: Grade 2 | 0
  Baseline: Erosion/Ulceration: Grade 3 | 0
  At Day 5: Erosion/Ulceration: number analyzed (Participants) | 101
  At Day 5: Erosion/Ulceration: Grade 0 | 97
  At Day 5: Erosion/Ulceration: Grade 1 | 4
  At Day 5: Erosion/Ulceration: Grade 2 | 0
  At Day 5: Erosion/Ulceration: Grade 3 | 0

2. Primary Outcome: Number of Participants Categorized by Local Tolerability Score by Visit for Each Individual Signs (Erythema, Flaking/Scaling, Crusting, Swelling, Vesiculation/Pustulation, and Erosion/Ulceration) at Day 8
Description: Local tolerability score was evaluated by investigator in terms of presence and absence of erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration signs and its severity in the areas of body where medication was applied. These symptoms were assessed by using a 4 - point grade scale of 0 - 3, where a score of 0=absent, 1=mild (slightly, barely perceptible), 2=moderate (distinct presence), and 3=severe (marked, intense). The higher score indicates severe symptoms. Number of participants categorized by local tolerability score by visit for each individual signs (erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration) at Day 8 were reported.
Time Frame: Baseline, Day 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tirbanibulin (Klisyri®)
Number analyzed (Participants) | 105
Participants
  Baseline: Erythema: Grade 0 | 81
  Baseline: Erythema: Grade 1 | 19
  Baseline: Erythema: Grade 2 | 5
  Baseline: Erythema: Grade 3 | 0
  At Day 8: Erythema: number analyzed (Participants) | 102
  At Day 8: Erythema: Grade 0 | 9
  At Day 8: Erythema: Grade 1 | 32
  At Day 8: Erythema: Grade 2 | 57
  At Day 8: Erythema: Grade 3 | 4
  Baseline: Flaking/Scaling: Grade 0 | 84
  Baseline: Flaking/Scaling: Grade 1 | 17
  Baseline: Flaking/Scaling: Grade 2 | 4
  Baseline: Flaking/Scaling: Grade 3 | 0
  At Day 8: Flaking/Scaling: number analyzed (Participants) | 102
  At Day 8: Flaking/Scaling: Grade 0 | 18
  At Day 8: Flaking/Scaling: Grade 1 | 43
  At Day 8: Flaking/Scaling: Grade 2 | 33
  At Day 8: Flaking/Scaling: Grade 3 | 8
  Baseline: Crusting: Grade 0 | 103
  Baseline: Crusting: Grade 1 | 2
  Baseline: Crusting: Grade 2 | 0
  Baseline: Crusting: Grade 3 | 0
  At Day 8: Crusting: number analyzed (Participants) | 102
  At Day 8: Crusting: Grade 0 | 66
  At Day 8: Crusting: Grade 1 | 28
  At Day 8: Crusting: Grade 2 | 8
  At Day 8: Crusting: Grade 3 | 0
  Baseline: Swelling: Grade 0 | 105
  Baseline: Swelling: Grade 1 | 0
  Baseline: Swelling: Grade 2 | 0
  Baseline: Swelling: Grade 3 | 0
  At Day 8: Swelling: number analyzed (Participants) | 102
  At Day 8: Swelling: Grade 0 | 75
  At Day 8: Swelling: Grade 1 | 19
  At Day 8: Swelling: Grade 2 | 8
  At Day 8: Swelling: Grade 3 | 0
  Baseline: Vesiculation/Pustulation: Grade 0 | 105
  Baseline: Vesiculation/Pustulation: Grade 1 | 0
  Baseline: Vesiculation/Pustulation: Grade 2 | 0
  Baseline: Vesiculation/Pustulation: Grade 3 | 0
  At Day 8: Vesiculation/Pustulation: number analyzed (Participants) | 102
  At Day 8: Vesiculation/Pustulation: Grade 0 | 101
  At Day 8: Vesiculation/Pustulation: Grade 1 | 1
  At Day 8: Vesiculation/Pustulation: Grade 2 | 0
  At Day 8: Vesiculation/Pustulation: Grade 3 | 0
  Baseline: Erosion/Ulceration: Grade 0 | 105
  Baseline: Erosion/Ulceration: Grade 1 | 0
  Baseline: Erosion/Ulceration: Grade 2 | 0
  Baseline: Erosion/Ulceration: Grade 3 | 0
  At Day 8: Erosion/Ulceration: number analyzed (Participants) | 102
  At Day 8: Erosion/Ulceration: Grade 0 | 91
  At Day 8: Erosion/Ulceration: Grade 1 | 8
  At Day 8: Erosion/Ulceration: Grade 2 | 3
  At Day 8: Erosion/Ulceration: Grade 3 | 0

3. Primary Outcome: Number of Participants Categorized by Local Tolerability Score by Visit for Each Individual Signs (Erythema, Flaking/Scaling, Crusting, Swelling, Vesiculation/Pustulation, and Erosion/Ulceration) at Day 15
Description: Local tolerability score was evaluated by investigator in terms of presence and absence of erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration signs and its severity in the areas of body where medication was applied. These symptoms were assessed by using a 4 - point grade scale of 0 - 3, where a score of 0=absent, 1=mild (slightly, barely perceptible), 2=moderate (distinct presence), and 3=severe (marked, intense). The higher score indicates severe symptoms. Number of participants categorized by local tolerability score by visit for each individual signs (erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration) at Day 15 were reported.
Time Frame: Baseline, Day 15
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tirbanibulin (Klisyri®)
Number analyzed (Participants) | 105
Participants
  Baseline: Erythema: Grade 0 | 81
  Baseline: Erythema: Grade 1 | 19
  Baseline: Erythema: Grade 2 | 5
  Baseline: Erythema: Grade 3 | 0
  At Day 15: Erythema: number analyzed (Participants) | 101
  At Day 15: Erythema: Grade 0 | 33
  At Day 15: Erythema: Grade 1 | 61
  At Day 15: Erythema: Grade 2 | 7
  At Day 15: Erythema: Grade 3 | 0
  Baseline: Flaking/Scaling: Grade 0 | 84
  Baseline: Flaking/Scaling: Grade 1 | 17
  Baseline: Flaking/Scaling: Grade 2 | 4
  Baseline: Flaking/Scaling: Grade 3 | 0
  At Day 15: Flaking/Scaling: number analyzed (Participants) | 101
  At Day 15: Flaking/Scaling: Grade 0 | 54
  At Day 15: Flaking/Scaling: Grade 1 | 33
  At Day 15: Flaking/Scaling: Grade 2 | 13
  At Day 15: Flaking/Scaling: Grade 3 | 1
  Baseline: Crusting: Grade 0 | 103
  Baseline: Crusting: Grade 1 | 2
  Baseline: Crusting: Grade 2 | 0
  Baseline: Crusting: Grade 3 | 0
  At Day 15: Crusting: number analyzed (Participants) | 101
  At Day 15: Crusting: Grade 0 | 86
  At Day 15: Crusting: Grade 1 | 12
  At Day 15: Crusting: Grade 2 | 3
  At Day 15: Crusting: Grade 3 | 0
  Baseline: Swelling: Grade 0 | 105
  Baseline: Swelling: Grade 1 | 0
  Baseline: Swelling: Grade 2 | 0
  Baseline: Swelling: Grade 3 | 0
  At Day 15: Swelling: number analyzed (Participants) | 101
  At Day 15: Swelling: Grade 0 | 96
  At Day 15: Swelling: Grade 1 | 4
  At Day 15: Swelling: Grade 2 | 1
  At Day 15: Swelling: Grade 3 | 0
  Baseline: Vesiculation/Pustulation: Grade 0 | 105
  Baseline: Vesiculation/Pustulation: Grade 1 | 0
  Baseline: Vesiculation/Pustulation: Grade 2 | 0
  Baseline: Vesiculation/Pustulation: Grade 3 | 0
  At Day 15: Vesiculation/Pustulation: number analyzed (Participants) | 101
  At Day 15: Vesiculation/Pustulation: Grade 0 | 101
  At Day 15: Vesiculation/Pustulation: Grade 1 | 0
  At Day 15: Vesiculation/Pustulation: Grade 2 | 0
  At Day 15: Vesiculation/Pustulation: Grade 3 | 0
  Baseline: Erosion/Ulceration: Grade 0 | 105
  Baseline: Erosion/Ulceration: Grade 1 | 0
  Baseline: Erosion/Ulceration: Grade 2 | 0
  Baseline: Erosion/Ulceration: Grade 3 | 0
  At Day 15: Erosion/Ulceration: number analyzed (Participants) | 101
  At Day 15: Erosion/Ulceration: Grade 0 | 100
  At Day 15: Erosion/Ulceration: Grade 1 | 0
  At Day 15: Erosion/Ulceration: Grade 2 | 1
  At Day 15: Erosion/Ulceration: Grade 3 | 0

4. Primary Outcome: Number of Participants Categorized by Local Tolerability Score by Visit for Each Individual Signs (Erythema, Flaking/Scaling, Crusting, Swelling, Vesiculation/Pustulation, and Erosion/Ulceration) at Day 29
Description: Local tolerability score was evaluated by investigator in terms of presence and absence of erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration signs and its severity in the areas of body where medication was applied. These symptoms were assessed by using a 4 - point grade scale of 0 - 3, where a score of 0=absent, 1=mild (slightly, barely perceptible), 2=moderate (distinct presence), and 3=severe (marked, intense). The higher score indicates severe symptoms. Number of participants categorized by local tolerability score by visit for each individual signs (erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration) at Day 29 were reported.
Time Frame: Baseline, Day 29
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tirbanibulin (Klisyri®)
Number analyzed (Participants) | 105
Participants
  Baseline: Erythema: Grade 0 | 81
  Baseline: Erythema: Grade 1 | 19
  Baseline: Erythema: Grade 2 | 5
  Baseline: Erythema: Grade 3 | 0
  At Day 29: Erythema: number analyzed (Participants) | 100
  At Day 29: Erythema: Grade 0 | 74
  At Day 29: Erythema: Grade 1 | 26
  At Day 29: Erythema: Grade 2 | 0
  At Day 29: Erythema: Grade 3 | 0
  Baseline: Flaking/Scaling: Grade 0 | 84
  Baseline: Flaking/Scaling: Grade 1 | 17
  Baseline: Flaking/Scaling: Grade 2 | 4
  Baseline: Flaking/Scaling: Grade 3 | 0
  At Day 29: Flaking/Scaling: number analyzed (Participants) | 100
  At Day 29: Flaking/Scaling: Grade 0 | 84
  At Day 29: Flaking/Scaling: Grade 1 | 16
  At Day 29: Flaking/Scaling: Grade 2 | 0
  At Day 29: Flaking/Scaling: Grade 3 | 0
  Baseline: Crusting: Grade 0 | 103
  Baseline: Crusting: Grade 1 | 2
  Baseline: Crusting: Grade 2 | 0
  Baseline: Crusting: Grade 3 | 0
  At Day 29: Crusting: number analyzed (Participants) | 100
  At Day 29: Crusting: Grade 0 | 97
  At Day 29: Crusting: Grade 1 | 3
  At Day 29: Crusting: Grade 2 | 0
  At Day 29: Crusting: Grade 3 | 0
  Baseline: Swelling: Grade 0 | 105
  Baseline: Swelling: Grade 1 | 0
  Baseline: Swelling: Grade 2 | 0
  Baseline: Swelling: Grade 3 | 0
  At Day 29: Swelling: number analyzed (Participants) | 100
  At Day 29: Swelling: Grade 0 | 98
  At Day 29: Swelling: Grade 1 | 2
  At Day 29: Swelling: Grade 2 | 0
  At Day 29: Swelling: Grade 3 | 0
  Baseline: Vesiculation/Pustulation: Grade 0 | 105
  Baseline: Vesiculation/Pustulation: Grade 1 | 0
  Baseline: Vesiculation/Pustulation: Grade 2 | 0
  Baseline: Vesiculation/Pustulation: Grade 3 | 0
  At Day 29: Vesiculation/Pustulation: number analyzed (Participants) | 100
  At Day 29: Vesiculation/Pustulation: Grade 0 | 100
  At Day 29: Vesiculation/Pustulation: Grade 1 | 0
  At Day 29: Vesiculation/Pustulation: Grade 2 | 0
  At Day 29: Vesiculation/Pustulation: Grade 3 | 0
  Baseline: Erosion/Ulceration: Grade 0 | 105
  Baseline: Erosion/Ulceration: Grade 1 | 0
  Baseline: Erosion/Ulceration: Grade 2 | 0
  Baseline: Erosion/Ulceration: Grade 3 | 0
  At Day 29: Erosion/Ulceration: number analyzed (Participants) | 100
  At Day 29: Erosion/Ulceration: Grade 0 | 100
  At Day 29: Erosion/Ulceration: Grade 1 | 0
  At Day 29: Erosion/Ulceration: Grade 2 | 0
  At Day 29: Erosion/Ulceration: Grade 3 | 0

5. Primary Outcome: Number of Participants Categorized by Local Tolerability Score by Visit for Each Individual Signs (Erythema, Flaking/Scaling, Crusting, Swelling, Vesiculation/Pustulation, and Erosion/Ulceration) at Day 57
Description: Local tolerability score was evaluated by investigator in terms of presence and absence of erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration signs and its severity in the areas of body where medication was applied. These symptoms were assessed by using a 4 - point grade scale of 0 - 3, where a score of 0=absent, 1=mild (slightly, barely perceptible), 2=moderate (distinct presence), and 3=severe (marked, intense). The higher score indicates severe symptoms. Number of participants categorized by local tolerability score by visit for each individual signs (erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration) at Day 57 were reported.
Time Frame: Baseline, Day 57
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tirbanibulin (Klisyri®)
Number analyzed (Participants) | 105
Participants
  Baseline: Erythema: Grade 0 | 81
  Baseline: Erythema: Grade 1 | 19
  Baseline: Erythema: Grade 2 | 5
  Baseline: Erythema: Grade 3 | 0
  At Day 57: Erythema: number analyzed (Participants) | 102
  At Day 57: Erythema: Grade 0 | 95
  At Day 57: Erythema: Grade 1 | 7
  At Day 57: Erythema: Grade 2 | 0
  At Day 57: Erythema: Grade 3 | 0
  Baseline: Flaking/Scaling: Grade 0 | 84
  Baseline: Flaking/Scaling: Grade 1 | 17
  Baseline: Flaking/Scaling: Grade 2 | 4
  Baseline: Flaking/Scaling: Grade 3 | 0
  At Day 57: Flaking/Scaling: number analyzed (Participants) | 102
  At Day 57: Flaking/Scaling: Grade 0 | 99
  At Day 57: Flaking/Scaling: Grade 1 | 3
  At Day 57: Flaking/Scaling: Grade 2 | 0
  At Day 57: Flaking/Scaling: Grade 3 | 0
  Baseline: Crusting: Grade 0 | 103
  Baseline: Crusting: Grade 1 | 2
  Baseline: Crusting: Grade 2 | 0
  Baseline: Crusting: Grade 3 | 0
  At Day 57: Crusting: number analyzed (Participants) | 102
  At Day 57: Crusting: Grade 0 | 102
  At Day 57: Crusting: Grade 1 | 0
  At Day 57: Crusting: Grade 2 | 0
  At Day 57: Crusting: Grade 3 | 0
  Baseline: Swelling: Grade 0 | 105
  Baseline: Swelling: Grade 1 | 0
  Baseline: Swelling: Grade 2 | 0
  Baseline: Swelling: Grade 3 | 0
  At Day 57: Swelling: number analyzed (Participants) | 102
  At Day 57: Swelling: Grade 0 | 102
  At Day 57: Swelling: Grade 1 | 0
  At Day 57: Swelling: Grade 2 | 0
  At Day 57: Swelling: Grade 3 | 0
  Baseline: Vesiculation/Pustulation: Grade 0 | 105
  Baseline: Vesiculation/Pustulation: Grade 1 | 0
  Baseline: Vesiculation/Pustulation: Grade 2 | 0
  Baseline: Vesiculation/Pustulation: Grade 3 | 0
  At Day 57: Vesiculation/Pustulation: number analyzed (Participants) | 102
  At Day 57: Vesiculation/Pustulation: Grade 0 | 102
  At Day 57: Vesiculation/Pustulation: Grade 1 | 0
  At Day 57: Vesiculation/Pustulation: Grade 2 | 0
  At Day 57: Vesiculation/Pustulation: Grade 3 | 0
  Baseline: Erosion/Ulceration: Grade 0 | 105
  Baseline: Erosion/Ulceration: Grade 1 | 0
  Baseline: Erosion/Ulceration: Grade 2 | 0
  Baseline: Erosion/Ulceration: Grade 3 | 0
  At Day 57: Erosion/Ulceration: number analyzed (Participants) | 102
  At Day 57: Erosion/Ulceration: Grade 0 | 102
  At Day 57: Erosion/Ulceration: Grade 1 | 0
  At Day 57: Erosion/Ulceration: Grade 2 | 0
  At Day 57: Erosion/Ulceration: Grade 3 | 0

6. Primary Outcome: Number of Participants With Maximum Local Tolerability Score Post-baseline for Each Individual Signs (Erythema, Flaking/Scaling, Crusting, Swelling, Vesiculation/Pustulation, and Erosion/Ulceration)
Description: Maximum local tolerability score post baseline was defined as the highest grade of any LSR reported at any post-baseline visits for a participant. Local tolerability score was assessed for signs erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration using a 4 - point grade scale of 0 - 3, where a score of 0=absent, 1=mild (slightly, barely perceptible), 2=moderate (distinct presence), and 3=severe (marked, intense). The higher score indicates severe symptoms. If a participant maximum individual sign local tolerability score stayed at 0 throughout the study, the participant was considered censored at last local tolerability score observation. Number of participants with maximum local tolerability score for each individual signs including erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration were reported.
Time Frame: Baseline, Maximum post-baseline (up to Day 57)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tirbanibulin (Klisyri®)
Number analyzed (Participants) | 105
Participants
  Baseline: Erythema: Grade 0 | 81
  Baseline: Erythema: Grade 1 | 19
  Baseline: Erythema: Grade 2 | 5
  Baseline: Erythema: Grade 3 | 0
  At Maximum post-baseline (up to Day 57): Erythema: number analyzed (Participants) | 103
  At Maximum post-baseline (up to Day 57): Erythema: Grade 0 | 4
  At Maximum post-baseline (up to Day 57): Erythema: Grade 1 | 27
  At Maximum post-baseline (up to Day 57): Erythema: Grade 2 | 66
  At Maximum post-baseline (up to Day 57): Erythema: Grade 3 | 6
  Baseline: Flaking/Scaling: Grade 0 | 84
  Baseline: Flaking/Scaling: Grade 1 | 17
  Baseline: Flaking/Scaling: Grade 2 | 4
  Baseline: Flaking/Scaling: Grade 3 | 0
  At Maximum post-baseline (up to Day 57): Flaking/Scaling: number analyzed (Participants) | 103
  At Maximum post-baseline (up to Day 57): Flaking/Scaling: Grade 0 | 16
  At Maximum post-baseline (up to Day 57): Flaking/Scaling: Grade 1 | 34
  At Maximum post-baseline (up to Day 57): Flaking/Scaling: Grade 2 | 44
  At Maximum post-baseline (up to Day 57): Flaking/Scaling: Grade 3 | 9
  Baseline: Crusting: Grade 0 | 103
  Baseline: Crusting: Grade 1 | 2
  Baseline: Crusting: Grade 2 | 0
  Baseline: Crusting: Grade 3 | 0
  At Maximum post-baseline (up to Day 57): Crusting: number analyzed (Participants) | 103
  At Maximum post-baseline (up to Day 57): Crusting: Grade 0 | 58
  At Maximum post-baseline (up to Day 57): Crusting: Grade 1 | 34
  At Maximum post-baseline (up to Day 57): Crusting: Grade 2 | 11
  At Maximum post-baseline (up to Day 57): Crusting: Grade 3 | 0
  Baseline: Swelling: Grade 0 | 105
  Baseline: Swelling: Grade 1 | 0
  Baseline: Swelling: Grade 2 | 0
  Baseline: Swelling: Grade 3 | 0
  At Maximum post-baseline (up to Day 57): Swelling: number analyzed (Participants) | 103
  At Maximum post-baseline (up to Day 57): Swelling: Grade 0 | 64
  At Maximum post-baseline (up to Day 57): Swelling: Grade 1 | 28
  At Maximum post-baseline (up to Day 57): Swelling: Grade 2 | 11
  At Maximum post-baseline (up to Day 57): Swelling: Grade 3 | 0
  Baseline: Vesiculation/Pustulation: Grade 0 | 105
  Baseline: Vesiculation/Pustulation: Grade 1 | 0
  Baseline: Vesiculation/Pustulation: Grade 2 | 0
  Baseline: Vesiculation/Pustulation: Grade 3 | 0
  At Maximum post-baseline (up to Day 57): Vesiculation/Pustulation: number analyzed (Participants) | 103
  At Maximum post-baseline (up to Day 57): Vesiculation/Pustulation: Grade 0 | 99
  At Maximum post-baseline (up to Day 57): Vesiculation/Pustulation: Grade 1 | 4
  At Maximum post-baseline (up to Day 57): Vesiculation/Pustulation: Grade 2 | 0
  At Maximum post-baseline (up to Day 57): Vesiculation/Pustulation: Grade 3 | 0
  Baseline: Erosion/Ulceration: Grade 0 | 105
  Baseline: Erosion/Ulceration: Grade 1 | 0
  Baseline: Erosion/Ulceration: Grade 2 | 0
  Baseline: Erosion/Ulceration: Grade 3 | 0
  At Maximum post-baseline (up to Day 57): Erosion/Ulceration: number analyzed (Participants) | 103
  At Maximum post-baseline (up to Day 57): Erosion/Ulceration: Grade 0 | 90
  At Maximum post-baseline (up to Day 57): Erosion/Ulceration: Grade 1 | 9
  At Maximum post-baseline (up to Day 57): Erosion/Ulceration: Grade 2 | 4
  At Maximum post-baseline (up to Day 57): Erosion/Ulceration: Grade 3 | 0

7. Primary Outcome: Time to Maximum Local Tolerability Score for Erythema, Flaking/Scaling, Crusting, Swelling, Vesiculation/Pustulation, and Erosion/Ulceration
Description: Time to maximum local tolerability score (in days) for each individual sign was calculated as [Date of first post-baseline occurrence of maximum local tolerability score for this individual sign - Date of first dose]. If a participant maximum individual sign LTA score stays at 0 throughout the study, the participants was considered censored at their last LTA score observation. Maximum local tolerability score was assessed for each signs using a 4 - point scale of 0 - 3, where 0 = absent, 1= mild, 2= moderate and 3 = severe. The higher score indicates severe symptoms. Time to maximum local tolerability score for erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration was reported.
Time Frame: Baseline up to Day 57
Population: The safety population included all enrolled participants who received at least 1 dose of the study drug. Here, "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies participants who were evaluable for specified categories.
Measure: Mean (Full Range); unit: Days
Arm/Group | Tirbanibulin (Klisyri®)
Number analyzed (Participants) | 99
Days
  Erythema | 4.0 [4 to 14]
  Flaking/Scaling: number analyzed (Participants) | 87
  Flaking/Scaling | 7.0 [4 to 15]
  Crusting: number analyzed (Participants) | 45
  Crusting | 7.0 [4 to 28]
  Swelling: number analyzed (Participants) | 39
  Swelling | 4.0 [4 to 12]
  Vesiculation/Pustulation: number analyzed (Participants) | 4
  Vesiculation/Pustulation | 4.0 [4 to 7]
  Erosion/Ulceration: number analyzed (Participants) | 13
  Erosion/Ulceration | 7.0 [4 to 14]

8. Primary Outcome: Local Tolerability Signs Total Composite Score by Visit at Day 5
Description: Local tolerability signs composite score by visit was defined as the sum of the scores graded from 0 (absent) to 3 (severe) on all six individual tolerability sign categories - erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration which gave total composite score ranged from 0 to 18. The higher score indicates severe symptoms. Local tolerability signs total composite score assessed from baseline up to Day 5 was reported.
Time Frame: Baseline, Day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tirbanibulin (Klisyri®)
Number analyzed (Participants) | 105
Score on a scale
  Baseline | 0.5 (1.06)
  At Day 5: number analyzed (Participants) | 101
  At Day 5 | 2.6 (1.67)

9. Primary Outcome: Local Tolerability Signs Total Composite Score by Visit at Day 8
Description: Local tolerability signs composite score by visit was defined as the sum of the scores graded from 0 (absent) to 3 (severe) on all six individual tolerability sign categories - erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration which gave total composite score ranged from 0 to 18. The higher score indicates severe symptoms. Local tolerability signs total composite score by visit at Day 8 was reported.
Time Frame: Baseline, Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Tirbanibulin (Klisyri®)
Number analyzed (Participants) | 105
Score on a Scale
  Baseline | 0.5 (1.06)
  At Day 8: number analyzed (Participants) | 102
  At Day 8 | 3.8 (2.25)

10. Primary Outcome: Local Tolerability Signs Total Composite Score by Visit at Day 15
Description: Local tolerability signs composite score by visit was defined as the sum of the scores graded from 0 (absent) to 3 (severe) on all six individual tolerability sign categories - erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration which gave total composite score ranged from 0 to 18. The higher score indicates severe symptoms. Local tolerability signs total composite score by visit at Day 15 was reported.
Time Frame: Baseline, Day 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Tirbanibulin (Klisyri®)
Number analyzed (Participants) | 105
Score on a Scale
  Baseline | 0.5 (1.06)
  At Day 15: number analyzed (Participants) | 101
  At Day 15 | 1.6 (1.46)

11. Primary Outcome: Local Tolerability Signs Total Composite Score by Visit at Day 29
Description: Local tolerability signs composite score by visit was defined as the sum of the scores graded from 0 (absent) to 3 (severe) on all six individual tolerability sign categories - erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration which gave total composite score ranged from 0 to 18. The higher score indicates severe symptoms. Local tolerability signs total composite score by visit at Day 29 was reported.
Time Frame: Baseline, Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Tirbanibulin (Klisyri®)
Number analyzed (Participants) | 105
Score on a Scale
  Baseline | 0.5 (1.06)
  At Day 29: number analyzed (Participants) | 100
  At Day 29 | 0.5 (0.80)

12. Primary Outcome: Local Tolerability Signs Total Composite Score by Visit at Day 57
Description: Local tolerability signs composite score by visit was defined as the sum of the scores graded from 0 (absent) to 3 (severe) on all six individual tolerability sign categories - erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration which gave total composite score ranged from 0 to 18. The higher score indicates severe symptoms. Local tolerability signs total composite score by visit at Day 57 was reported.
Time Frame: Baseline, Day 57
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Tirbanibulin (Klisyri®)
Number analyzed (Participants) | 105
Score on a Scale
  Baseline | 0.5 (1.06)
  At Day 57: number analyzed (Participants) | 102
  At Day 57 | 0.1 (0.36)

13. Primary Outcome: Maximum Local Tolerability Signs Total Composite Score Post Baseline
Description: The maximum local tolerability signs composite score across visits was derived as the maximum local tolerability composite score observed post-baseline. Local tolerability signs composite score was defined as the sum of the scores graded from 0 (absent) to 3 (severe) on all six individual tolerability sign categories - erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration which gave total composite score ranged from 0 to 18. The higher score indicates severe symptoms. Maximum local tolerability signs total composite score post baseline was reported.
Time Frame: Baseline, Maximum post-baseline (up to Day 57)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tirbanibulin (Klisyri®)
Number analyzed (Participants) | 105
Score on a scale
  Baseline | 0.5 (1.06)
  At Maximum post-baseline (up to Day 57): number analyzed (Participants) | 103
  At Maximum post-baseline (up to Day 57) | 4.1 (2.12)

14. Primary Outcome: Time to Maximum Local Tolerability Total Composite Score
Description: Time to maximum composite local tolerability score (in days) was calculated as (Date of first post-baseline occurrence of maximum composite local tolerability score - Date of first dose). The maximum local tolerability signs composite score across visits was derived as the maximum local tolerability composite score observed post-baseline. Local tolerability signs composite score was defined as the sum of the scores graded from 0 (absent) to 3 (severe) on all six individual tolerability sign categories - erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration which gave total composite score ranged from 0 to 18. The higher score indicates severe symptoms. If a participant's maximum composite local tolerability score stays at 0 throughout the study, the participant was considered censored at their last local tolerability score observation. Time to maximum local tolerability total composite score was reported.
Time Frame: Baseline up to Day 57
Population: The safety population included all enrolled participants who received at least 1 dose of the study drug. Here, "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tirbanibulin (Klisyri®)
Number analyzed (Participants) | 100
Days | 7.0 [6.01 to 7.31]

15. Primary Outcome: Number of Participants With Pigmentation and Scarring in the Treatment Area by Visit at Day 5
Description: Absence and presence of pigmentation (i.e., hypopigmentation and hyperpigmentation) and scarring in the treatment field by visit at Day 5 was reported.
Time Frame: Baseline, Day 5
Population: The safety population included all enrolled participants who received at least 1 dose of the study drug. Here, "number analyzed" signifies participants who were evaluable for specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Tirbanibulin (Klisyri®)
Number analyzed (Participants) | 105
Participants
  Baseline: Hypopigmentation Presence | 22
  Baseline: Hypopigmentation Absence | 83
  At Day 5: Hypopigmentation Presence: number analyzed (Participants) | 100
  At Day 5: Hypopigmentation Presence | 22
  At Day 5: Hypopigmentation Absence: number analyzed (Participants) | 100
  At Day 5: Hypopigmentation Absence | 78
  Baseline: Hyperpigmentation Presence | 28
  Baseline: Hyperpigmentation Absence | 77
  At Day 5: Hyperpigmentation Presence: number analyzed (Participants) | 100
  At Day 5: Hyperpigmentation Presence | 26
  At Day 5: Hyperpigmentation Absence: number analyzed (Participants) | 100
  At Day 5: Hyperpigmentation Absence | 74
  Baseline: Scarring Presence | 12
  Baseline: Scarring Absence | 93
  At Day 5: Scarring Presence: number analyzed (Participants) | 100
  At Day 5: Scarring Presence | 12
  At Day 5: Scarring Absence: number analyzed (Participants) | 100
  At Day 5: Scarring Absence | 88

16. Primary Outcome: Number of Participants With Pigmentation and Scarring in the Treatment Area by Visit at Day 8
Description: Absence and presence of pigmentation (i.e., hypopigmentation and hyperpigmentation) and scarring in the treatment field by visit at Day 8 was reported.
Time Frame: Baseline, Day 8
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Tirbanibulin (Klisyri®)
Number analyzed (Participants) | 105
Participants
  Baseline: Hypopigmentation Presence | 22
  Baseline: Hypopigmentation Absence | 83
  At Day 8: Hypopigmentation Presence: number analyzed (Participants) | 101
  At Day 8: Hypopigmentation Presence | 21
  At Day 8: Hypopigmentation Absence: number analyzed (Participants) | 101
  At Day 8: Hypopigmentation Absence | 80
  Baseline: Hyperpigmentation Presence | 28
  Baseline: Hyperpigmentation Absence | 77
  At Day 8: Hyperpigmentation Presence: number analyzed (Participants) | 101
  At Day 8: Hyperpigmentation Presence | 23
  At Day 8: Hyperpigmentation Absence: number analyzed (Participants) | 101
  At Day 8: Hyperpigmentation Absence | 78
  Baseline: Scarring Presence | 12
  Baseline: Scarring Absence | 93
  At Day 8: Scarring Presence: number analyzed (Participants) | 101
  At Day 8: Scarring Presence | 13
  At Day 8: Scarring Absence: number analyzed (Participants) | 101
  At Day 8: Scarring Absence | 88

17. Primary Outcome: Number of Participants With Pigmentation and Scarring in the Treatment Area by Visit at Day 15
Description: Absence and presence of pigmentation (i.e., hypopigmentation and hyperpigmentation) and scarring in the treatment field by visit at Day 15 was reported.
Time Frame: Baseline, Day 15
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Tirbanibulin (Klisyri®)
Number analyzed (Participants) | 105
Participants
  Baseline: Hypopigmentation Presence | 22
  Baseline: Hypopigmentation Absence | 83
  At Day 15: Hypopigmentation Presence: number analyzed (Participants) | 101
  At Day 15: Hypopigmentation Presence | 21
  At Day 15: Hypopigmentation Absence: number analyzed (Participants) | 101
  At Day 15: Hypopigmentation Absence | 80
  Baseline: Hyperpigmentation Presence | 28
  Baseline: Hyperpigmentation Absence | 77
  At Day 15: Hyperpigmentation Presence: number analyzed (Participants) | 101
  At Day 15: Hyperpigmentation Presence | 20
  At Day 15: Hyperpigmentation Absence: number analyzed (Participants) | 101
  At Day 15: Hyperpigmentation Absence | 81
  Baseline: Scarring Presence | 12
  Baseline: Scarring Absence | 93
  At Day 15: Scarring Presence: number analyzed (Participants) | 101
  At Day 15: Scarring Presence | 11
  At Day 15: Scarring Absence: number analyzed (Participants) | 101
  At Day 15: Scarring Absence | 90

18. Primary Outcome: Number of Participants With Pigmentation and Scarring in the Treatment Area by Visit at Day 29
Description: Absence and presence of pigmentation (i.e., hypopigmentation and hyperpigmentation) and scarring in the treatment field by visit at Day 29 was reported.
Time Frame: Baseline, Day 29
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Tirbanibulin (Klisyri®)
Number analyzed (Participants) | 105
Participants
  Baseline: Hypopigmentation Presence | 22
  Baseline: Hypopigmentation Absence | 83
  At Day 29: Hypopigmentation Presence: number analyzed (Participants) | 100
  At Day 29: Hypopigmentation Presence | 20
  At Day 29: Hypopigmentation Absence: number analyzed (Participants) | 100
  At Day 29: Hypopigmentation Absence | 80
  Baseline: Hyperpigmentation Presence | 28
  Baseline: Hyperpigmentation Absence | 77
  At Day 29: Hyperpigmentation Presence: number analyzed (Participants) | 100
  At Day 29: Hyperpigmentation Presence | 16
  At Day 29: Hyperpigmentation Absence: number analyzed (Participants) | 100
  At Day 29: Hyperpigmentation Absence | 84
  Baseline: Scarring Presence | 12
  Baseline: Scarring Absence | 93
  At Day 29: Scarring Presence: number analyzed (Participants) | 100
  At Day 29: Scarring Presence | 10
  At Day 29: Scarring Absence: number analyzed (Participants) | 100
  At Day 29: Scarring Absence | 90

19. Primary Outcome: Number of Participants With Pigmentation and Scarring in the Treatment Area by Visit at Day 57
Description: Absence and presence of pigmentation (i.e., hypopigmentation and hyperpigmentation) and scarring in the treatment field by visit at Day 57 was reported.
Time Frame: Baseline, Day 57
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Tirbanibulin (Klisyri®)
Number analyzed (Participants) | 105
Participants
  Baseline: Hypopigmentation Presence | 22
  Baseline: Hypopigmentation Absence | 83
  At Day 57: Hypopigmentation Presence: number analyzed (Participants) | 102
  At Day 57: Hypopigmentation Presence | 18
  At Day 57: Hypopigmentation Absence: number analyzed (Participants) | 102
  At Day 57: Hypopigmentation Absence | 84
  Baseline: Hyperpigmentation Presence | 28
  Baseline: Hyperpigmentation Absence | 77
  At Day 57: Hyperpigmentation Presence: number analyzed (Participants) | 102
  At Day 57: Hyperpigmentation Presence | 16
  At Day 57: Hyperpigmentation Absence: number analyzed (Participants) | 102
  At Day 57: Hyperpigmentation Absence | 86
  Baseline: Scarring Presence | 12
  Baseline: Scarring Absence | 93
  At Day 57: Scarring Presence: number analyzed (Participants) | 102
  At Day 57: Scarring Presence | 9
  At Day 57: Scarring Absence: number analyzed (Participants) | 102
  At Day 57: Scarring Absence | 93

20. Primary Outcome: Number of Participants With Any Treatment-emergent Adverse Events (TEAEs), Serious TEAEs and Adverse Events of Special Interest (AESIs)
Description: TEAEs were defined as either those adverse events (AEs) with an onset after dosing or those pre-existing conditions that worsened after dosing. An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered an Investigational Product. An SAE with any untoward medical occurrence that at any dose, resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect in the child of a participant who was exposed to the study drug, or any other medically important event that may jeopardize the patient or require intervention to prevent one of the other outcomes. AESI's included in this study were skin cancers (including basal cell carcinoma, squamous cell carcinoma, and melanoma) based on their relevance for the current intended use. TEAEs included both serious and non-serious AEs.
Time Frame: Baseline up to Day 57
Population: The safety population included all enrolled participants who received at least 1 dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Tirbanibulin (Klisyri®)
Number analyzed (Participants) | 105
Participants
  Participants with TEAEs | 29
  Participants with Serious TEAEs | 2
  Participants with AESIs | 2

21. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Laboratory Parameters
Description: Laboratory parameters included blood chemistry, hamatology, and urinalysis. Clinically significant laboratory abnormalities assessment was based on Investigator interpretation. Number of participants with clinically significant abnormalities in laboratory parameters (included hematology, blood chemistry and urinalysis) were reported.
Time Frame: Baseline up to Day 57
Population: The safety population included all enrolled participants who received at least 1 dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Tirbanibulin (Klisyri®)
Number analyzed (Participants) | 105
Participants | 0

22. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Vital signs included measurement of pulse rate, systolic and diastolic blood pressure, respiratory rate, and body temperature. Clinically significant vital signs abnormalities assessment was based on Investigator interpretation. Number of participants with clinically significant abnormalities in vital signs were reported.
Time Frame: Baseline up to Day 57
Population: The safety population included all enrolled participants who received at least 1 dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Tirbanibulin (Klisyri®)
Number analyzed (Participants) | 105
Participants | 1

23. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Physical Examination
Description: Physical examination included weight and height measurements. Clinically significant physical examination abnormalities assessment was based on Investigator interpretation. Number of participants with clinically significant abnormalities in physical examination were reported.
Time Frame: Baseline up to Day 57
Population: The safety population included all enrolled participants who received at least 1 dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Tirbanibulin (Klisyri®)
Number analyzed (Participants) | 105
Participants | 1

24. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Electrocardiogram (ECG)
Description: ECG included heart rhythm, heart rate, QRS intervals, QT intervals, RR intervals and corrected QT (QTc) intervals parameters measurement. Clinically significant ECGs abnormalities assessment was based on Investigator interpretation. Number of participants with clinically significant abnormalities in ECG were reported.
Time Frame: Baseline up to Day 57
Population: The safety population included all enrolled participants who received at least 1 dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Tirbanibulin (Klisyri®)
Number analyzed (Participants) | 105
Participants | 1

ADVERSE EVENTS:
Time Frame: Baseline up to Day 57
Description: The safety population included all enrolled participants who received at least 1 dose of the study drug.
Arm/Group | Tirbanibulin (Klisyri®)
All-Cause Mortality (participants affected / at risk) | 1/105
Serious Adverse Events (participants affected / at risk) | 2/105
Other Adverse Events (participants affected / at risk) | 29/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tirbanibulin (Klisyri®) (N=105)
Tachycardia (Cardiac disorders) | 1
Asthenia (General disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Encephalopathy (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tirbanibulin (Klisyri®) (N=105)
Atrial fibrillation (Cardiac disorders) | 1
Application site pruritus (General disorders) | 11
Application site pain (General disorders) | 9
Application site bruise (General disorders) | 1
Application site dryness (General disorders) | 1
Application site hypoaesthesia (General disorders) | 1
Oedema peripheral (General disorders) | 1
Tenderness (General disorders) | 1
Bronchitis (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Laryngitis viral (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT05279131/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/31/NCT05279131/SAP_001.pdf